CLINICAL TRIAL: NCT03612570
Title: Evaluation of Nano-Pulse Stimulation (NPS) in Sebaceous Hyperplasia
Brief Title: Nano-Pulse Stimulation (NPS) in Sebaceous Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-SH-006
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Skin Lesion; Skin Abnormalities; Sebaceous Hyperplasia
Keywords: Nano-Pulse Stimulation; NPS
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- NPS Treated SH Lesion (Experimental): Nano-Pulse Stimulation Device using pre-defined energy protocol
  Interventions: Device: Nano-Pulse Stimulation Device

INTERVENTIONS:
Device: Nano-Pulse Stimulation Device — NPS utilizes a timed series of low energy, high voltage nanosecond (billionth of a second) pulses which are applied directly to targeted tissue using small microneedles. NPS energy induces cell signaling and the activation of cellular pathways by creating transient nanopores in cellular membranes and organelles and initiate regulated cell death.

SUMMARY:
This prospective, open label, muti-center study evaluates the use of Nano-Pulse Stimulation (NPS) in the treatment of Sebaceous Hyperplasia (SH) lesions less than 2.5mm in size.

DETAILED DESCRIPTION:
The study is designed with each subject serving as his or her own control. A total of up to 75 subjects with 2-5 qualifying SH lesions will be enrolled and treated with either a 1.5-mm x 1.5-mm or 2.5-mm x 2.5-mm tip. All treated lesions will receive at least one NPS treatment and evaluated at 30 days for lesion clearance. Initial lesions scored as Not Clear or Partially Clear may undergo a second NPS treatment. All subjects will have their lesions evaluated at 60 days post-primary or secondary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Presents with at least 2 and up to 5 clinically visible SH lesions
* Understands that 1 lesion will remain untreated to act as a reference
* Lesions must measure no greater than 2.5 x 2.5 at the outside margin
* Wishes to have at least 1 and perhaps 2 NPS treatments to each study lesion
* Selection of the non-treated reference lesion will be randomly identified
* Willing to return for 4 or 5 total study visits at specified intervals over 60 or 90 days
* Agrees to photographic or other image capture methods of both the treated and untreated lesions.
* Agrees to avoid any other treatment to the NPS treated and untreated SH lesions until the end of the NPS study
* Has no evidence of active infection in the designated tissue prior to treatment and reports no infection within 90 days
* Is not allergic to Lidocaine or Lidocaine-like products

Exclusion Criteria:

* Presence of Implantable electronic devices that cannot be removed. e.g., pacemaker or automatic defibrillator
* Taking medications prescribed for cardiac arrhythmia at any time within 6 months prior to exposure to the NPS device
* SH lesions are located within the eye orbit or on the nose
* Active infection or history of infection in designated test area within 90 days prior to study initiation
* Use of oral steroid and/or retinoid use within the last 12 months
* Prior treatment to the identified SH lesions targeted for the study which occurred within 6 months prior to study start
* Is known to be immune-compromised and/or received immunosuppressant therapy within 6 months prior to study start
* Taking blood thinning medications
* Has Insulin dependent diabetes
* Is known to be pregnant or lactating female

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (5):
- United States (5):
  - Laser & Skin Surgery Medical Group, Inc., Sacramento, California
  - Premier Plastic Surgery, San Mateo, California
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialists, Edina, Minnesota
  - Dermatology, Laser & Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munavalli GS, Zelickson BD, Selim MM, Kilmer SL, Rohrer TE, Newman J, Jauregui L, Knape WA, Ebbers E, Uecker D, Nuccitelli R. Safety and Efficacy of Nanosecond Pulsed Electric Field Treatment of Sebaceous Gland Hyperplasia. Dermatol Surg. 2020 Jun;46(6):803-809. doi: 10.1097/DSS.0000000000002154. PMID 31592824

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: SH Lesions
Groups:
- Number of Study Participants: Total Number of Participants with Sebaceous Hyperplastic Lesions treated with Nano-Pulse Stimulation (NPS) using a pre-defined energy protocol.
Period: Overall Study
Arm/Group | Number of Study Participants
Started | 72; 226 SH Lesions
Completed | 71; 222 SH Lesions
Not Completed | 1; 4 SH Lesions
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: One Participant was not seen at follow-up after being treated or enrolled into the study.
Groups:
- All Participants: Nano-Pulse Stimulation Device using pre-defined energy protocol
  Nano-Pulse Stimulation Device: NPS utilizes a timed series of low energy, high voltage nanosecond (billionth of a second) pulses which are applied directly to targeted tissue using small microneedles. NPS energy induces cell signaling and the activation of cellular pathways by creating transient nanopores in cellular membranes and organelles and initiate regulated cell death.
Arm/Group | All Participants
Number analyzed (Participants) | 72
Age, Continuous [Mean (Full Range); unit: Years] | 55 [31 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Cleared SH Lesions
Description: SH lesion clearance was assessed live by investigators for each treated SH lesion (n=222) at 60-days post-last treatment using a 4-point scale (i.e., 0, 1, 2, 3) where each number corresponded to Clear, Mostly Clear, Partially Clear, or Not Clear, respectively. Lower scores mean better outcome, i.e., 0=Clear while a 3=Not Clear.
Time Frame: 60-days follow-up post-last treatment
Population: Total number of treated SH Lesions at 60-days.
Measure: Number; unit: Percentage of cleared SH Lesions
Units Other Than Participants: SH lesions
Groups:
- Total Number of Cleared Lesions With Sebaceous Hyperplasia (SH): Total Number of Lesions with Sebaceous Hyperplasia (SH) that were treated with Nano-Pulse Stimulation (NPS) using a pre-defined energy protocol
Arm/Group | Total Number of Cleared Lesions With Sebaceous Hyperplasia (SH)
Number analyzed (Participants) | 71
Number analyzed (SH lesions) | 222
Percentage of cleared SH Lesions | 99.5

ADVERSE EVENTS:
Time Frame: Skin effects (hyperpigmentation) were observed per SH lesion at the 5-day, 30-day, 60-day and if applicable 90-day follow-up periods.
Description: Skin effects per SH lesion were defined as presence of mild, moderate or severe post-inflammatory hyperpigmentation (PIH).
Groups:
- NPS Treated Sebaceous Hyperplasia (SH) Lesion: Nano-Pulse Stimulation (NPS) treated SH Lesions using pre-defined treatment levels. All adverse events were recorded per lesion.
Arm/Group | NPS Treated Sebaceous Hyperplasia (SH) Lesion
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 32/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPS Treated Sebaceous Hyperplasia (SH) Lesion (N=71)
Post-Inflammatory Hyperpigmentation (Skin and subcutaneous tissue disorders) | 32 (32) — Transient PIH per lesion (n=222) at 60-days post-NPS treatment was 45% with Mild (32%, n=70), Moderate (10%, n=23), Moderate to Severe (2%, n=5) and Severe (1%, n=3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03612570/Prot_003.pdf